CLINICAL TRIAL: NCT03726047
Title: Feedback and Cognition During Locomotor Learning Post Stroke
Brief Title: Exercise and Motor Learning After Stroke (Study #3)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1139080-3
Record Dates: First submitted 2018-10-30; First posted 2018-10-31 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Subjects will complete learning of a new walking pattern through distorted visual feedback and retention will be tested immediately after and 24 hours later (without visual feedback).
- Exercise (Experimental): Subjects will complete learning of a new walking pattern through distorted visual feedback and retention will be tested immediately without visual feedback. This will be followed immediately by 5 minutes of high intensity exercise. Retention without visual feedback will them be tested again 24 hours later.
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Subjects will complete 5 minutes of exercise on an ergometer to examine the effects of exercise on retention of a newly learned walking pattern.
  Arms: Exercise

SUMMARY:
Subjects with chronic stroke (> 6 months post-stroke) will learn a new walking pattern through distorted visual feedback. Retention of the pattern will be tested without visual feedback immediately after learning and 24 hours later. Subjects will be randomly assigned to the control group or the exercise group. The control group will simply complete the learning task. The exercise group will complete 5 minutes of exercise immediately following the first retention test to test for the effects of exercise on retention 24 hours later.

DETAILED DESCRIPTION:
Despite significant time and money spent on post-stroke rehabilitation, stroke survivors are left with reduced walking capacity and significant disability. After stroke, individuals must relearn movements that have been disrupted due to damage to the brain, therefore, enhancing motor learning is critical to improving the rehabilitation of walking after stroke. In this project investigators will examine how individual factors influence motor learning after stroke and use this information to personalize post-stroke rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

Age 18-85 Single, unilateral, chronic stroke (>6 months post-stroke), confirmed by MRI or CT scan Score >1 on question 1b and >0 on question 1c of the NIH Stroke Scale Able to walk at self-selected speed without assistance from another person Resting heart rate between 40-100 beats per minute Resting blood pressure between 90/60 to 185/100

Exclusion Criteria:

Evidence of cerebellar stroke on clinical MRI or CT scan, because of role of cerebellum in learning Other neurologic conditions in addition to stroke Inability to walk outside the home prior to the stroke Coronary artery bypass graft or myocardial infarction within past 3 months, Musculoskeletal pain that limits walking Inability to communicate with investigators Visual field cut Neglect Unexplained dizziness in last 6 months

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
24 hour retention | 24 hours
  This is amount of learning that was retained when subjects return 24 hours later and are tested without visual feedback

CONTACTS AND LOCATIONS:
Overall Officials: Darcy Reisman, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thompson ED, Bhat S, French MA, Morton S, Pohlig RT, Reisman DS. Effects of an Acute High Intensity Exercise Bout on Retention of Explicit, Strategic Locomotor Learning in Individuals With Chronic Stroke. Neurorehabil Neural Repair. 2023 Sep;37(9):628-639. doi: 10.1177/15459683231195039. Epub 2023 Aug 30. PMID 37646138